CLINICAL TRIAL: NCT04953546
Title: Clinical Application of the Apex of the Deep Cartilage in Evaluating the Position of the Femoral Tunnel of the Anterior Cruciate Ligament Reconstruction
Brief Title: Clinical Application of the Apex of the Deep Cartilage in Evaluating the Femoral Tunnel of the ACL Reconstruction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2021212
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: anterior cruciate ligament; computed tomography; the apex of the deep cartilage; microscopic evaluation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ACL group: According to the previous clinical diagnosis, volunteers who has suffered the ACL injury.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is an observation study, with no intervention

SUMMARY:
With the apex of the deep cartilage (ADC) as the symbol, the consistency of the two methods in the postoperatively computed tomography (CT) and microscopic evaluation of the position of the femoral tract of the anterior cruciate ligament (ACL) was studied.Expected results:P1 and P2, D1 and D2 were positively correlated, and the linear relationship was significant. Bland-Altman diagram shows a good consistency.

DETAILED DESCRIPTION:
Objectives:

With the apex of the deep cartilage (ADC) as the symbol, the consistency of the two methods in the postoperatively computed tomography (CT) and microscopic evaluation of the position of the femoral tract of the anterior cruciate ligament (ACL) was studied.

Methods:

Prospective cohort study.

Fifty-two patients requiring arthroscopic anterior cruciate ligament reconstruction were enrolled in the Sports Medicine Department of Peking University Third Hospital.

Collect patients' basic information and preoperative conditions. During the operation, the patient's knee was bent 90°, and the center point was positioned according to the intact femoral stump. The horizontal distance from the ADC to the anterior bone margin (L1) and the horizontal distance from the center point of the bone tract (L1) were measured by the master, the first aid and the second aid, and the distance from the center point of the bone tract to the lower bone margin (D1) was measured, and the ratio of L1 /L1 was calculated (P1).

The horizontal distance from the ADC to the anterior bone margin (L2) and the horizontal distance from the center of the bone tract (L2) were measured by three investigators on postoperative CT films, and the distance from the center of the bone tract to the lower bone margin (D2) was also measured, and the ratio of L2 /L2 was calculated (P2).

Linear regression, Pearson correlation and Bland-Altman analysis were used to compare the consistency between the endoscopic assessment and CT assessment.

Expected results:

P1 and P2, D1 and D2 were positively correlated, and the linear relationship was significant. Bland-Altman diagram shows a good consistency.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have isolated ACL injury and receive ACL reconstruction surgery at Peking University Third Hospital.
* With isolated ACL injury (an ACL injury with no need for surgical repairs to other knee structures).
* All participants have no known disorders or diseases other than ACL rupture.

Exclusion Criteria:

• Other injuries affecting movement performance.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inclusion Criteria: Patients who have isolated ACL injury and receive ACL reconstruction surgery at Peking University Third Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
The horizontal distance from the ADC to the anterior bone margin | On the 1 day of enrollment.
  The patients were measured microscopically at the time of surgery and again on CT after surgery.
the horizontal distance from the center point of the bone tract | On the 1 day of enrollment.
  The patients were measured microscopically at the time of surgery and again on CT
the distance from the center point of the bone tract to the lower bone margin | On the 1 day of enrollment.
  The patients were measured microscopically at the time of surgery and again on CT

CONTACTS AND LOCATIONS:
Overall Officials: Yong Ma, Doctor, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No